CLINICAL TRIAL: NCT01062750
Title: Liver Regeneration Therapy by Intrahepatic Arterial Administration of Autologous Adipose Tissue Derived Stromal Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanazawa University (Other)
Responsible Party: Principal Investigator, Shuichi Kaneko, Professor, Kanazawa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1132
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adipose tissue derived stromal cells (Other)
  Interventions: Biological: adipose tissue derived stromal cells dosage

INTERVENTIONS:
Biological: adipose tissue derived stromal cells dosage — single administration of autologous adipose tissue derived stroma cells via intrahepatic arterial catheterization

SUMMARY:
Mesenchymal stem cells have capability to differentiate into hepatocyte and will be useful for liver regeneration. Adipose tissue is relatively enriched with mesenchymal stem cell compared to bone marrow tissue. In this trial, eligible liver cirrhosis patients will receive autologous adipose tissue derived stromal cells through intrahepatic arterial catheterization.

DETAILED DESCRIPTION:
The population of the liver cirrhosis patients is enormous in Japan and the only radical treatment for them is liver transplantation: however, the number of giving donor is extremely limited. Mesenchymal stem cells have been capable to differentiate into mesodermal-lineage cells as well as endodermal-lineage cells such as hepatocytes. They reside in the mesenchymal tissues such as bone marrows as well as adipose tissues. The latter tissues are relatively enriched with mesenchymal stem cells compared to bone marrow cells. In this study, the cirrhotic patients will undergo intrahepatic arterial administration of autologous adipose tissue derived stromal cells through catheter.

ELIGIBILITY:
Criteria defined in the implementation protocol

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
all cause harmful events | one month

CONTACTS AND LOCATIONS:
Overall Officials: Shuichi Kaneko, M.D., Study Chair — Kanazawa University
Locations (1):
- Kanazawa University Hospital, Kanazawa, Ishikawa-ken, Japan